CLINICAL TRIAL: NCT00008528
Title: A Phase III Open-Label, Randomized, Active-Controlled Study Assessing the Efficacy and Safety of T-20 (HIV-1 Fusion Inhibitor) in Combination With an Optimized Background Regimen, Versus Optimized Background Therapy Alone, in Patients With Prior Experience and/or Prior Documented Resistance to Each of the Three Classes of Approved Antiretrovirals (Nucleoside Reverse Transcriptase, Non-Nucleoside Reverse Transcriptase and Protease Inhibitors)
Brief Title: T-20 With Anti-HIV Combination Therapy for Patients With Prior Anti-HIV Drug Treatment and/or Drug Resistance to Each of the Three Classes of Approved Anti-HIV Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trimeris (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 295C; T20-301
Record Dates: First submitted 2001-01-12; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-06

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Drug Resistance, Microbial; RNA, Viral; Membrane Fusion; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

INTERVENTIONS:
Drug: Enfuvirtide

SUMMARY:
The purpose of this study is to compare the change in viral load (amount of HIV in the blood) of patients who receive T-20 with selected anti-HIV drugs to that of patients who receive only selected anti-HIV drugs.

DETAILED DESCRIPTION:
Eligible patients remain on their pre-study regimen until baseline. An OB regimen is chosen by the physician and patient based on the patient's prior treatment history, prior and current laboratory abnormalities, the screening GT/PT antiretroviral resistance testing, and any prior GT/PT antiretroviral resistance (if available). The drugs in the OB regimen are chosen from among the currently approved antiretrovirals and permitted newly approved/investigational antiretrovirals available in the countries where the study is implemented, and must consist of 3 to 5 drugs, including no more than 1 newly approved/investigational agent. Patients are stratified with respect to viral load and use (versus non-use) of any of the allowed newly approved/investigational antiretrovirals. Patients are randomized to receive 1 of the following 2 treatments for 48 weeks: OB or OB plus T-20. Patients are followed to assess viral load, safety, antiretroviral resistance, T-20 pharmacokinetics, and quality of life. At the end of 48 weeks of treatment patients are allowed to (a) roll over and receive OB plus T-20 (for patients receiving OB regimen alone) or (b) continue taking OB plus T-20 (for patients already receiving OB plus T-20), for an additional 48 weeks (plus 4 weeks safety follow-up period), or until 12 weeks after commercial availability of T-20 in the country in which they are treated, whichever comes first. All patients are followed in this study for a maximum of 100 weeks from their initial baseline visit date.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-infected.
* Are at least 16 years old (have consent of parent or guardian if under 18).
* Have a viral load (level of HIV in the blood) of 5,000 copies/ml or more.
* Have received anti-HIV drugs for at least 6 months and/or have shown resistance to each of the 3 types of anti-HIV drugs as follows: nucleoside reverse transcriptase inhibitors (resistant to 1 or more); nonnucleoside reverse transcriptase inhibitors (resistant to 1 or more); and protease inhibitors (resistant to 2 or more, taken either together or 1 after the other for at least 6 months total).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 525

CONTACTS AND LOCATIONS:
Locations (37):
- United States (34):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Body Positive, Phoenix, Arizona
  - Pacific Oaks Med Group, Beverly Hills, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Univ of California, San Diego, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - San Francisco VA Med Ctr, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Whitman Walker Clinic/Elizabeth Taylor Med Ctr, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Steinhart Medical Associates, Miami, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Trevor Slom, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - New England Med Ctr, Boston, Massachusetts
  - Massachusetts Gen Hosp, Boston, Massachusetts
  - Community Research Initiative of New England, Brookline, Massachusetts
  - Regions Hosp, Saint Paul, Minnesota
  - Albany Med College, Albany, New York
  - Peter Tsang, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of North Carolina / SOCA, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ / AIDS Clinical Trials Unit, Cleveland, Ohio
  - Oregon Health Sciences Univ, Portland, Oregon
  - MCP Hahnemann Univ, Philadelphia, Pennsylvania
  - Pennsylvania Oncology and Hematology Associates, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Nicholas Bellos, Dallas, Texas
  - Univ of Texas Med Branch, Galveston, Texas
  - Univ of Texas / Thomas Street Clinic, Houston, Texas
  - Univ of Washington / AIDS Clinical Trial Unit, Seattle, Washington
  - Vancouver Clinic, Vancouver, Washington
- Canada (3):
  - Toronto Gen Hosp, Toronto, Ontario
  - Centre Hospitalier de la Universite de Montreal (CHUM), Montreal, Quebec
  - Clinique Medicale L'Actuele, Montreal, Quebec

REFERENCES:
- [Background] Lalezari JP, Henry K, O'Hearn M, Montaner JS, Piliero PJ, Trottier B, Walmsley S, Cohen C, Kuritzkes DR, Eron JJ Jr, Chung J, DeMasi R, Donatacci L, Drobnes C, Delehanty J, Salgo M; TORO 1 Study Group. Enfuvirtide, an HIV-1 fusion inhibitor, for drug-resistant HIV infection in North and South America. N Engl J Med. 2003 May 29;348(22):2175-85. doi: 10.1056/NEJMoa035026. Epub 2003 Mar 13. PMID 12637625